CLINICAL TRIAL: NCT03409198
Title: A Randomized Phase IIb Study Evaluating Immunogenic Chemotherapy Combined with Ipilimumab and Nivolumab in Patients with Metastatic Hormone Reseptor Positive Breast Cancer
Brief Title: Phase IIb Study Evaluating Immunogenic Chemotherapy Combined with Ipilimumab and Nivolumab in Breast Cancer
Acronym: ICON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry); Helse Stavanger HF (Other Government); Helse Sor-Ost (Other Government); Sorlandet Hospital HF (Other Government); Jules Bordet Institute (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Centre Hospitalier Universitaire UCLouvain Namur (Other)
Responsible Party: Principal Investigator, Jon Amund Kyte, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICON CA209-9FN
Record Dates: First submitted 2017-12-04; First posted 2018-01-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Hormone Receptor Positive Tumor; Metastatic Breast Cancer
Keywords: Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Ipilimumab; Nivolumab; liposomal doxorubicin; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Randomized, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): Chemo only (pegylated liposomal doxorubicin + cyclophosphamide)
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Cyclophosphamide
- Arm B (Experimental): Chemo + ipilimumab + nivolumab
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Pegylated liposomal doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab blocks CTLA-4 and may deplete regulatory T cells
  Other Names: Yervoy
  Arms: Arm B
Drug: Nivolumab — Nivolumab blocks PD-1 and thereby enhances the effector phase of the immune reaction, by enabling T cells to kill tumor cells and engage effectively with other PD-L1 expressing targets.
  Other Names: Opdivo
  Arms: Arm B
Drug: Pegylated liposomal doxorubicin — Chemotherapy
Drug: Cyclophosphamide — Chemotherapy

SUMMARY:
Breast cancer is rarely curable after metastasis, and the therapeutic options are limited. Interestingly, the host immune response is strongly predictive for the effect of chemotherapy in subgroups of patients with breast cancer. The aim is to release the brake on the immune response by use of ipilimumab, which blocks CTLA-4 and may deplete regulatory T cells, combined with nivolumab (anti PD1). Importantly, it is possible that non-responders to nivolumab/ipilimumab (nivo/ipi) can be turned responders by use of immunogenic chemotherapy.

DETAILED DESCRIPTION:
There is compelling evidence from animal studies, supported by data from humans, that some chemotherapeutic agents are immunogenic. Doxorubicin and cyclophosphamide have been shown to be particularly powerful inducers of immunogenic cell death. Both agents fulfil 5/5 criteria established for assessing the immunogenicity of different chemotherapeutic drugs. There is also strong evidence from humans, particularly in breast cancer, indicating that the clinical effect of doxorubicin and cyclophosphamide depends on the host immune response. Further, these agents have been shown to induce a Type I interferon immune response in breast cancer. Taken together, there is a strong rationale for synergy between doxorubicin/cyclophosphamide and PD-1/CTLA-4 blockade. The trial combines nivolumab and ipilimumab with established 1st choice chemotherapy in patients with metastatic hormone reseptor positive breast cancer. Nivolumab/ipilimumab (nivo/ipi) may i) potentiate the patient´s spontaneous anti-tumor immune response ii) synergize with chemotherapeutic agents that induce immunological cell death

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic hormone receptor positive breast cancer (primary or recurrent), defined as ER+ >1% in metastatic biopsy (archival material or study biopsy) or cytology and HER2 negative in the last biopsy or cytology evaluable for HER2. HER2-analysis is to be perfomed according to national criteria.
2. Adequate core or excisional study biopsy of a tumor lesion. Lesions in previously irradiated areas may only be used for the biopsy if the lesion has appared or progressed after radiation. No anti-tumor treatment is allowed between the time point for biopsy and study entry.
3. Measurable metastatic disease according to RECIST
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Signed Informed Consent Form
6. Women or men aged ≥ 18 years
7. A minimum of 12 months from adjuvant/neoadjuvant chemotherapy with antracyclins to relapse disease
8. A maximum of one previous line with chemotherapy in the metastatic setting
9. Chemotherapy is considered as preferred treatment
10. Previous endocrine and targeted therapy is allowed
11. No use of systemic corticosteroids at study entry
12. Female subject of childbearing potential should have a negative urine or serum pregnancy within 7 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
13. Female subjects of childbearing potential should agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year, during the treatment period and for at least 5 months after the last dose of study therapy.
14. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy
15. Able to swallow and retain orally administered medication
16. Adequate organ function as defined in Table 1

Exclusion Criteria:

1. Malignancies other than breast cancer within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer)
2. Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 8 weeks prior to randomization
3. Known CNS disease, except for asymptomatic CNS metastases, provided all of the following criteria are met:

   1. Measurable disease outside the CNS
   2. Asymptomatic for CNS disease > 4 weeks
   3. No ongoing requirement for corticosteroids as therapy for CNS disease
   4. No radiation of brain lesions within 2 weeks prior to randomization
   5. No leptomeningeal disease
4. Uncontrolled pleural effusion, pericardial effusion, or ascites. Patients with indwelling catheters (e.g., PleurX®) are allowed
5. Uncontrolled tumor-related pain. Patients requiring narcotic pain medication must be on a stable regimen at study entry. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to randomization. Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not presently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to randomization
6. Ionized calcium > 1.2 x UNL. The use of bisphosphonates is allowed
7. Pregnant or breastfeeding
8. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome)
9. Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within 3 months prior to randomization, unstable arrhythmias, or unstable angina Patients with a known left ventricular ejection fraction (LVEF) < 40% will be excluded. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
10. Severe infection within 21 days prior to randomization, requiring hospitalization
11. Received oral or IV antibiotics within 1 week prior to Cycle 1, Day 1. Patients receiving routine antibiotic prophylaxis (e.g., to prevent chronic obstructive pulmonary disease exacerbation or for dental extraction) are eligible
12. Major surgical procedure within 21 days prior to randomization or anticipation of the need for a major surgical procedure during the course of the study other than for diagnosis. Placement of central venous access catheter(s) is not considered a major surgical procedure and is therefore permitted
13. A history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
14. Known hypersensitivity to any of the components of the investigational products
15. A history of autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxin, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only (e.g., no psoriatic arthritis) are permitted provided that they meet all of the following conditions:

    1. Rash must cover less than 10% of body surface area.
    2. Disease is well controlled at baseline and only requiring low potency topical steroids
    3. No acute exacerbations of underlying condition within the last 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids)
16. Undergone allogeneic stem cell or solid organ transplantation
17. A history of idiopathic pulmonary fibrosis pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
18. A positive test for HIV
19. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
20. Active tuberculosis
21. Currently receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
22. Received treatment with immune checkpoint modulators, including anti-CTLA-4, anti-PD-1, or anti-PD-L1 therapeutic antibodies
23. Received treatment with systemic immunostimulatory agents (including but not limited to interferons or IL-2) within 4 weeks or five half-lives of the drug (whichever is shorter) prior to randomization
24. Received treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to randomization, or anticipated requirement for systemic immunosuppressive medications during the trial

    1. Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study
    2. Patients with a history of allergic reaction to IV contrast requiring steroid pre-treatment should have baseline and subsequent tumor assessments performed using MRI
    3. The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed
25. Received anti-cancer therapy (medical agents or radiation) within 2 weeks prior to study Cycle 1, Day 1. Palliative radiotherapy for bone lesions is allowed up to 7 days before start of therapy.
26. A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator
27. Known psychiatric or substance abuse disorders that would interfere with cooperation and the requirements of the trial
28. Received a live vaccine within 30 days of planned start of study therapy, or is expected to receive such a vaccine while on therapy

    a. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
29. Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-01-21 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Toxicity: CTCAE v4.0 | 3 years
  Assessment of toxicity of combined treatment with ipilimumab, nivolumab, pegylated liposomal doxorubicin and cyclophosphamide (ipi/nivo/chemo)
Progression-free survival (PFS) | We expect to reach the data-driven time point for PFS-analysis (95% PFS in the control group) approximately 3 years after the study opens. If this is not met within 24 months after inclusion of the last patient, the PFS-analysis will be performed at this
  Assessment of clinical response in ipi/nivo/chemo group compared to chemo only group: Progression-free survival (PFS); compare the PFS rates when 95% of patients in the control croup have PD

SECONDARY OUTCOMES:
Duration of Response (DR) | 3 years
  Assessment of clinical response in ipi/nivo/chemo group compared to chemo only group: duration of response (DR)
Overall Survival (OS) | 5 years
  Assessment of clinical response in ipi/nivo/chemo group compared to chemo only group: overall survival (OS)
Duration of Response (DR) in cross-over arm | 3 years
  Assessment of clinical response in ipi/nivo group: duration of response (DR)
Overall Suvival (OS) in cross-over arm | 5 years
  Assessment of clinical response in ipi/nivo group: overall survival (OS)
Toxicity, cross-over arm, CTCAE v4.0 | 3 years
  Assessment of toxicity of ipi/nivo (without chemotherapy) in cross-over arm
Objective tumor Response Rate (ORR) | 3 years
  Assessment of clinical response in ipi/nivo/chemo group compared to chemo only group: Objective tumor response rate (ORR)
Durable tumor Response Rate (DRR) | 3 years
  Assessment of clinical response in ipi/nivo/chemo group compared to chemo only group: durable tumor response rate (DRR; >6 months)
Objective tumor Response Rate (ORR) in cross-over arm | 3 years
  Assessment of clinical response in ipi/nivo group: Objective tumor response rate (ORR)
Durable tumor Response Rate (DRR) in cross-over arm | 3 years
  Assessment of clinical response in ipi/nivo group: durable tumor response rate (DRR; >6 months)
Clinical Benefit Rate (CBR) | 3 years
  Proportion of patients with an objective tumor response or with stable disease lasting at least 6 months
Clinical Benefit Rate (CBR) in cross-over arm | 3 years
  Proportion of patients with an objective tumor response or with stable disease lasting at least 6 months
PD-L1 expression | 3 years
  Assessment of PD-L1 expression, mutation load and immune gene expression as biomarkers for clinical response
Chalder Fatigue Questionnaire (FQ) | 3 years
  Assessment of patient reported outcomes, as measured by the Chalder Fatigue Questionnaire (FQ)
Pain intensity | 3 years
  Assessment of patient reported outcomes, as measured by an 11 point Numerical Rating Scale (NRS) for pain intensity
EORTC QLQ-C15-PAL | 3 years
  Assessment of patient reported outcomes, as measured by the EORTC QLQ-C15-PAL
Biological response in molecular subtypes of breast cancer | 3 years
  Comparison of clinical and biological response in molecular subtypes of breast cancer

OTHER OUTCOMES:
Immunological response | 3 years
  Assessment of immunological response. In selected patients, the specificity of T-cell responses will be analysed. The analysis will be based neoantigen prediction and will be performed by multimer technology.
Biomarkers for clinical response | 3 years
  Identification of biomarkers for clinical response by use of gene profiling, pathology, cytokine assays and other analysis on material from study patients. The following predefined biomarkers will be compared between responders and non-responders: PD-L1 in biopsies, immune gene signature in biopsies. Further explorative investigations will be performed to identify new candidate biomarker signatures.
Biomarkers for toxicity | 3 years
  Identification of biomarkers for toxicity by use of gene profiling, pathology, cytokine assays and other analysis on material from study patients. The analysis is explorative and will be performed to identify new candidate biomarker signatures. The candidate signatures will be compared between patients with and without immune related adverse events.
Assessment of changes in the immunological milieu in tumor and peripheral blood | 3 years
  Considering each study arm separately, and by comparing arm A to arm B. The assessment will be performed by flow cytometry and CyTOF of immune cells, and by gene expression profiling of tumor biopsies. In periferal blood,the frequency of immune cell subsets will be determined and compared between baseline and later timepoints. In biopsies, gene expression profiles will be compared between baseline and later timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Amund Kyte, Principal Investigator — Oslo University Hospital
Locations (6):
- Belgium (3):
  - Institut Jules Bordet, Brussels, Brussels Capital
  - Cliniques universitaires Saint-Luc, Brussels, Brussels Capital
  - CHU UCL Namur, Namur, Namur
- Norway (3):
  - Soerlandet Hospital HF Kristiansand, Kristiansand
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andresen NK, Rossevold AH, Quaghebeur C, Gilje B, Boge B, Gombos A, Falk RS, Mathiesen RR, Julsrud L, Garred O, Russnes HG, Lereim RR, Chauhan SK, Lingjaerde OC, Dunn C, Naume B, Kyte JA. Ipilimumab and nivolumab combined with anthracycline-based chemotherapy in metastatic hormone receptor-positive breast cancer: a randomized phase 2b trial. J Immunother Cancer. 2024 Jan 19;12(1):e007990. doi: 10.1136/jitc-2023-007990. PMID 38242720
- [Derived] Kyte JA, Andresen NK, Russnes HG, Fretland SO, Falk RS, Lingjaerde OC, Naume B. ICON: a randomized phase IIb study evaluating immunogenic chemotherapy combined with ipilimumab and nivolumab in patients with metastatic hormone receptor positive breast cancer. J Transl Med. 2020 Jul 3;18(1):269. doi: 10.1186/s12967-020-02421-w. PMID 32620163